CLINICAL TRIAL: NCT05251337
Title: Use of Aromatherapy to Reduce Symptom Burden in Patients Receiving Stem Cell Transplantation
Brief Title: Use of Aromatherapy to Reduce Symptom Burden
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: Indiana University Health (Other)
Responsible Party: Principal Investigator, Monica Bates, Registered Nurse, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 11973
Record Dates: First submitted 2022-02-03; First posted 2022-02-22 (Actual); Results first posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-04

CONDITIONS: Anxiety; Chemotherapy-induced Nausea and Vomiting
Keywords: stem cell transplant; anxiety; chemotherapy-induced nausea and vomiting; aromatherapy
MeSH Terms: conditions — Anxiety Disorders; Vomiting | interventions — Oils, Volatile

STUDY DESIGN:
Intervention Model Description: Prior to randomization, participants will be asked which symptom, nausea/vomiting or anxiety, is most burdensome for them. Participants will be stratified based on their identified symptom of burden (nausea/vomiting or anxiety) and will then be randomized to either the intervention or control group, with a target of 50 participants in the nausea/vomiting symptom group (25 intervention and 25 control) and 50 participants in the anxiety symptom group (25 intervention and 25 control).
Who Masked: Participant
Masking Description: Participants will not be informed of assignment to intervention or control; however, the blank aromatherapy patch (control group) will not have a scent and the essential oil infused aromatherapy patch (intervention group) will. Thus, it may be obvious to participants what group they are randomized to.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Intervention - nausea/vomiting (Experimental): Patients indicating that nausea/vomiting is their primary symptom of concern and are randomized to receive intervention will be allocated to the intervention - nausea/vomiting arm. This arm will receive peppermint inhaled aromatherapy patches (or mandarin as an alternative if they have a peppermint sensitivity).
  Interventions: Drug: Essential oils
- Intervention - anxiety (Experimental): Patients indicating that anxiety is their primary symptom of concern and are randomized to receive intervention will be allocated to the intervention - anxiety arm. This arm will receive lavender inhaled aromatherapy patches.
  Interventions: Drug: Essential oils
- Control - nausea/vomiting (Placebo Comparator): Patients indicating that nausea/vomiting is their primary symptom of concern and are randomized to receive control will be allocated to the control - nausea/vomiting arm. This arm will receive blank (no essential oil infusion) aromatherapy patches.
  Interventions: Drug: Placebo
- Control - anxiety (Placebo Comparator): Patients indicating that anxiety is their primary symptom of concern and are randomized to receive control will be allocated to the control - anxiety arm. This arm will receive blank (no essential oil infusion) aromatherapy patches.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Essential oils — Participants will receive Wyndmere Naturals, Inc. aromatherapy patches. The hydrogel adhesive patches are infused with essential oil for inhaled aromatherapy treatment. The aromatherapy patches provide an occlusive barrier that is hypoallergenic, allowing essential oils to be inhaled without coming in direct contact with the skin. Participants indicating nausea/vomiting is their symptom of concern will receive peppermint aromatherapy patches (or mandarin if peppermint sensitivity). Participants indicating anxiety is their symptom of concern will receive lavender aromatherapy patches.
  Arms: Intervention - anxiety; Intervention - nausea/vomiting
Drug: Placebo — Patients assigned to either control group (nausea/vomiting or anxiety) will receive Wyndmere Naturals non-scented patches (i.e., blank hydrogel adhesive patches without essential oil infusion).
  Arms: Control - anxiety; Control - nausea/vomiting

SUMMARY:
The purpose of this study is to evaluate the effect of inhaled aromatherapy on symptoms of nausea/vomiting and anxiety in patients who have received a stem cell transplant. Aromatherapy involves essential oils from aromatic plants that can be absorbed into the body in different ways. Our study will be using inhaled aromatherapy, which has been found helpful for symptoms such as nausea/vomiting and anxiety.

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the efficacy of aromatherapy on symptoms of chemotherapy-induced nausea, vomiting, and retching (CINVR) and anxiety for patients hospitalized for hematopoietic stem cell transplant. The primary aim will be to evaluate the effect of inhaled aromatherapy on CINVR and anxiety symptoms compared to control for 48 hours. Secondary aims include (1) Evaluating patient satisfaction with aromatherapy at completion of study; (2) Evaluating the antiemetic administration between intervention and control groups during the 48-hour intervention time span; (3) Evaluating the number and incidence of unit falls pre and post intervention.

This study will be a randomized controlled trial. Prior to randomization, participants will be asked which symptom, nausea/vomiting or anxiety, is most burdensome for them. Participants will be stratified based on their identified symptom of burden (nausea/vomiting or anxiety) and will then be randomized to either the intervention or control group, with a target of 50 participants in the nausea/vomiting symptom group (25 intervention and 25 control) and 50 participants in the anxiety symptom group (25 intervention and 25 control). Intervention and control groups will receive Wyndmere Naturals, Inc. aromatherapy patches and a symptom diary. Participants in the intervention group indicating that nausea/vomiting is the primary symptom of concern will receive peppermint inhaled aromatherapy patches (or mandarin if peppermint intolerance indicted). Participants in the intervention group indicating that anxiety is the primary symptoms of concern with receive lavender inhaled aromatherapy patches. The control group will receive non-scented aromatherapy patches (i.e., blank hydrogel adhesive patches without essential oil infusion), so it will not be feasible to blind participants to group assignment. The control group will have the same interactions with the study team as the intervention group and will complete patch changes and a symptom diary to serve as an attention control.

ELIGIBILITY:
Inclusion Criteria:

* Patients from a bone marrow transplant unit or hematology/oncology unit within an adult academic health center in the Midwest.
* Adult stem cell transplant inpatients that have received autologous or allogeneic transplant and are actively going through therapy.
* Patients must also be alert and oriented, able to interact with the study team, and able to read and write English.

Exclusion Criteria:

* Under 18 years of age
* Intubation
* Medical sedation
* Receipt of chimeric antigen receptor T (CAR-T) cells
* History of atrial fibrillation
* History of seizures/epilepsy
* Adhesive allergy or sensitivity
* Currently pregnant
* Prisoner

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 92 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-06-22 (Actual); Study Completion 2023-06-22 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Indiana University Health, University Hospital, Indianapolis, Indiana, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Intervention - Nausea/Vomiting | Intervention - Anxiety | Control - Nausea/Vomiting | Control - Anxiety
Started | 24 | 21 | 26 | 21
Completed | 19 | 15 | 20 | 17
Not Completed | 5 | 6 | 6 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention - Nausea/Vomiting | Intervention - Anxiety | Control - Nausea/Vomiting | Control - Anxiety | Total
Number analyzed (Participants) | 24 | 21 | 26 | 21 | 92
Age, Continuous [Mean (Full Range); unit: Years] | 55 [22 to 72] | 51 [24 to 79] | 52 [22 to 78] | 51 [21 to 70] | 52 [21 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 16 | 10 | 12 | 55
  Male | 7 | 5 | 16 | 9 | 37
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Native American or American Indian | 0 | 0 | 0 | 0 | 0
  Asian or Pacific Islander | 0 | 0 | 1 | 0 | 1
  Latino | 0 | 1 | 0 | 0 | 1
  Black or African American | 4 | 3 | 3 | 2 | 12
  White/Non-Hispanic | 20 | 17 | 22 | 19 | 78
  Other | 0 | 0 | 0 | 0 | 0
  Prefer Not to Say | 0 | 0 | 0 | 0 | 0
Transplant Type [Count of Participants; unit: Participants]
  Allogenic | 1 | 3 | 5 | 7 | 16
  Autologous | 23 | 18 | 21 | 14 | 76
Cancer Type [Count of Participants; unit: Participants]
  Leukemia | 1 | 3 | 4 | 4 | 12
  Dendritic Cell | 0 | 0 | 1 | 0 | 1
  Germ Cell Tumor | 3 | 2 | 4 | 1 | 10
  Hodgkin's Disease | 0 | 3 | 0 | 3 | 6
  Myelodysplastic Syndromes | 0 | 0 | 0 | 2 | 2
  Multiple Myeloma | 20 | 13 | 16 | 11 | 60
  Non-Hodgkin's Lymphoma | 0 | 0 | 1 | 0 | 1
Chemotherapy Regimen [Count of Participants; unit: Participants]
  BEAM | 0 | 3 | 1 | 2 | 6
  Etoposide/Carboplatin | 3 | 2 | 4 | 1 | 10
  Fludarabine/Cytoxan/Total Body Irradiation | 0 | 0 | 1 | 0 | 1
  Fludarabine/Cytoxan | 0 | 0 | 1 | 3 | 4
  Melphalan | 20 | 13 | 16 | 11 | 60
  Thiotepa/Cytoxan | 1 | 3 | 2 | 4 | 10
  Triptycene/Cytoxan/Fludarabine | 0 | 0 | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Chemotherapy-induced Nausea, Vomiting, and Retching (CINVR) Symptoms at Baseline, 25 Hours, and 48 Hours
Description: CINVR involves three gastrointestinal symptoms (nausea, vomiting, retching) influenced by administration of chemotherapy. Nausea is expressed as an unpleasant feeling in the throat/epigastrium that can result in expulsion of stomach content, known as vomiting. Retching is the effort to expel stomach contents without success. The Rhodes Index of Nausea, Vomiting and Retching (INVR) was used to measure CINVR and includes 8 Likert-type items on a 5-point scale. Items are scored from 0 (least amount of distress) to 4 (the most distress) and added after reverse coding items 1,3,6, and 7 to calculate an overall INVR score. The overall score ranges from 0 to 32, with higher scores indicating higher symptom burden. Subscales for symptom experience, occurrence, and distress for each symptom (nausea, vomiting, retching) are calculated by adding corresponding scale items for each subscale. The ranges for each subscale were as follows: nausea experience (0-12), vomiting experience (0-12),
Time Frame: baseline (0 hours) and post-intervention (24, 48 hours)
Population: Outcome measure was pre-specified to analyze data only from the "Intervention-Nausea/Vomiting" and "Control-Nausea/Vomiting" Arms
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Nausea/Vomiting | Control - Nausea/Vomiting
Number analyzed (Participants) | 24 | 26
score on a scale
  Baseline | 9.6 (4.6) | 8.5 (4.4)
  24 hours | 5.2 (3.1) | 4.9 (3.5)
  48 hours | 3.9 (3.5) | 4.4 (4.4)
Statistical Analysis 1: Comparison: Intervention - Nausea/Vomiting vs Control - Nausea/Vomiting; Test type: Superiority; p = 0.462, Mixed Models Analysis

2. Primary Outcome: Anxiety Symptoms at Baseline 24 Hours, and 48 Hours
Description: Anxiety is defined as excessive or persistent worry about aspects of life. Anxiety was measured using a shortened version of Spielberger's State Anxiety Inventory (SAI). The original SAI contains 20 items to measure state anxiety and items are scored using a 4-point Likert-type scale (almost never-almost always). The shortened SAI retains 6 items (from the original 20) and has evidence supporting good internal reliability consistency and strong construct validity. Items are scored from 1 (not at all) to 4 (very much so) and added after reverse coding anxiety absent items, with higher total scores indicating higher state anxiety. The shortened SAI total score ranges from a total score of 6-24.
Time Frame: baseline (0 hours) and post-intervention (24, 48 hours)
Population: Outcome measure was pre-specified to analyze data only from the "Intervention-Anxiety" and "Control-Anxiety" Arms/Groups
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Intervention - Anxiety | Control - Anxiety
Number analyzed (Participants) | 21 | 21
score on a scale
  Baseline | 14.4 (3.7) | 15.4 (4.1)
  24 hours | 10.9 (3.3) | 13.3 (3.5)
  48 hours | 10.5 (3.4) | 12.9 (4.1)
Statistical Analysis 1: Comparison: Intervention - Anxiety vs Control - Anxiety; Test type: Superiority; p = 0.285, Mixed Models Analysis

3. Secondary Outcome: Patient Satisfaction at 48 Hours
Description: An investigator-developed questionnaire was administered at the 48-hour study completion to evaluate patient satisfaction. Participants rated their satisfaction with the intervention on a 1-10 rating scale, with 10 being extremely satisfied (e.g., higher score means higher satisfaction).
Time Frame: post-intervention (48 hours)
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention - Nausea/Vomiting | Intervention - Anxiety | Control - Nausea/Vomiting | Control - Anxiety
Number analyzed (Participants) | 21 | 15 | 20 | 18
Participants
  Rating = 1 | 0 | 0 | 0 | 0
  Rating = 2 | 0 | 0 | 1 | 0
  Rating = 3 | 0 | 0 | 2 | 0
  Rating = 4 | 0 | 0 | 1 | 0
  Rating = 5 | 0 | 2 | 2 | 1
  Rating = 6 | 1 | 1 | 3 | 5
  Rating = 7 | 2 | 0 | 3 | 0
  Rating = 8 | 5 | 3 | 5 | 2
  Rating = 9 | 8 | 2 | 1 | 4
  Rating =10 | 5 | 7 | 2 | 6

4. Secondary Outcome: Medications Administered for Nausea/Vomiting Indication for 48 Hour Study Timeframe
Description: Medications administered for nausea/vomiting indication (scopolamine, lorazepam, promethazine, prochlorperazine, olanzapine, dexamethasone, Marinol, ondansetron). Medications administered for nausea/vomiting symptom indication were extracted from the electronic medical record for participants in the nausea/vomiting symptom group.
Time Frame: 48 hour intervention timeframe
Population: Outcome measure was pre-specified to collect data only from the "Intervention-Nausea/Vomiting" and "Control-Nausea/Vomiting" Arms/Groups
Measure: Mean (Standard Deviation); unit: Medications Administered
Arm/Group | Intervention - Nausea/Vomiting | Control - Nausea/Vomiting
Number analyzed (Participants) | 24 | 26
Medications Administered | 10.0 (5.0) | 7.1 (5.3)
Statistical Analysis 1: Comparison: Intervention - Nausea/Vomiting vs Control - Nausea/Vomiting; Test type: Superiority; p = 0.091, t-test, 2 sided

5. Secondary Outcome: Inpatient Fall Events at Baseline and During Intervention
Description: Fall numbers using total number of falls reported to the National Database of Nurse Quality Indicators. Data were extracted from the bone marrow transplant and hematology/oncology units for baseline (December 2020-March 2022) and intervention (March 2022-June 2023) timeframes.
Time Frame: baseline (December 2020-February 2022) and during intervention (March 2022-June 2023)
Population: Data were pre-specified to be analyzed across participating hospital units, rather than study arms.
Measure: Number; unit: Fall Events
Units Other Than Participants: Hospital Units
Groups:
- Participating Units: Bone marrow transplant unit and hematology/oncology unit within an adult academic health center in Midwest
Arm/Group | Participating Units
Number analyzed (Participants) | 2
Number analyzed (Hospital Units) | 2
Fall Events
  Baseline | 32
  Post | 31

ADVERSE EVENTS:
Time Frame: Events monitored from enrollment to 72 hours post enrollment for intervention group participants only (control did not receive essential oils).
Description: Adverse Event Definition Per Study Protocol: Any problematic medical occurrence/changes in medical condition, regardless of causality, in a study participant who received the intervention from enrollment - 72 hours post.
  Adverse events were not monitored for "Control-Nausea/Vomiting" or "Control-Anxiety" Arms/Groups.
Groups:
- Intervention - Nausea/Vomiting: Participants indicating that nausea/vomiting was their primary symptom of concern and were randomized to receive intervention were allocated to the intervention - nausea/vomiting arm. This arm received peppermint inhaled aromatherapy patches (or mandarin as an alternative if they had a peppermint sensitivity).
- Intervention - Anxiety: Participants indicating that anxiety was their primary symptom of concern and were randomized to receive intervention were allocated to the intervention - anxiety arm. This arm received lavender inhaled aromatherapy patches.
Arm/Group | Intervention - Nausea/Vomiting | Intervention - Anxiety
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21
Serious Adverse Events (participants affected / at risk) | 0/24 | 1/21
Other Adverse Events (participants affected / at risk) | 9/24 | 12/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention - Nausea/Vomiting (N=24) | Intervention - Anxiety (N=21)
Sepsis (Infections and infestations) | 0 (0) | 1 (1) — Not related
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) — Not related
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention - Nausea/Vomiting (N=24) | Intervention - Anxiety (N=21)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) — Possibly related
Dysuria (Renal and urinary disorders) | 0 (0) | 3 (3) — Not related
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 2 (2) — Unlikely related
Abdominal Cramps (Gastrointestinal disorders) | 2 (2) | 0 (0) — Unlikely related
Headache (Nervous system disorders) | 2 (2) | 2 (2) — Possibly related
Hypokalemia (Metabolism and nutrition disorders) | 2 (2) | 0 (0) — Unlikely related
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1)
Vomiting (Gastrointestinal disorders) | 3 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 5 (5) | 4 (4)
Mucositis (Infections and infestations) | 6 (6) | 3 (3)
Fatigue (General disorders) | 3 (3) | 6 (6)
Neutropenic Fever (Immune system disorders) | 5 (5) | 3 (3)
Pancytopenia (Immune system disorders) | 6 (6) | 4 (4)
Orthostasis (General disorders) | 3 (3) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-08-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT05251337/Prot_SAP_001.pdf